CLINICAL TRIAL: NCT02947711
Title: An Open-label, Single-Sequence, Drug-Drug Interaction Study to Evaluate the Effect of Diltiazem Extended Release on the Pharmacokinetics of E2027 in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Diltiazem Extended Release on the Pharmacokinetics of E2027 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2027-A001-003
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Healthy Subjects
Keywords: E2027; Healthy participants; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E2027 100 mg alone and in combination with diltiazem ER 300 mg (Experimental): E2027 100 milligrams (mg) will be administered orally on Days 1 and 12. Diltiazem extended release (ER) 300 mg will be administered alone on Days 7 to 24; however, on the morning of Day 12 it will be coadministered with E2027 100 mg.
  Interventions: Drug: E2027; Drug: Diltiazem ER

INTERVENTIONS:
Drug: E2027 — 2 x 50 mg capsules, once daily on Day 1 and Day 12
Drug: Diltiazem ER — 1 x 300 mg capsule, once daily on Days 7 through 24

SUMMARY:
This Phase 1, open-label, single-sequence, drug-drug Interaction study is conducted to evaluate the effect of diltiazem extended release (ER) (a moderate CYP3A inhibitor and P glycoprotein [Pgp] inhibitor) on the pharmacokinetics (PK) of a single oral dose of E2027 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, male or female participants, ≥18 years old and ≤50 years old at the time of informed consent
* Body mass index of 18 to 32 kilograms per meters squared (kg/m^2) at Screening

Exclusion Criteria:

* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks prior to the first dose
* Females who are: (a) breastfeeding; or (b) pregnant at Screening or Baseline (documented by a negative beta human chorionic gonadotropin [β-hCG] (or human chorionic gonadotropin [hCG]) test with a sensitivity of at least 25 International Units per Liter (IU/L) or equivalent units of β-hCG [or hCG]). Note: A negative urine pregnancy test is required before the administration of the first dose.
* Females of childbearing potential who:

  * Had unprotected sexual intercourse within 30 days before study entry and do not agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double barrier method [such as condom plus diaphragm with spermicide] or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 28 days after study drug discontinuation. Note: Hormonal contraceptives are not allowed.
  * Are currently (for at least 30 days) abstinent, and do not agree to use a double barrier method (as described above) or refrain from sexual activity during the study period or for 28 days after study drug discontinuation NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month prior to first dose).
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period or for 28 days after study drug discontinuation.
* Evidence of disease that may influence the outcome of the study within 4 weeks prior to the first dose (e.g., psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism)
* Any history of abdominal surgery that may affect pharmacokinetic profiles of E2027 (e.g., hepatectomy, nephrectomy, digestive organ resection). Participants with a history cholecystectomy or appendectomy are not excluded.
* Any other clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, electrocardiogram (ECG) finding (including a PR greater than 210 milliseconds (msec), a QRS greater than 110 msec), or laboratory test results that requires medical treatment at Screening or Baseline as determined by the Principal Investigator or designee
* A prolonged QT/QTc interval (QTc greater than 450 msec) demonstrated on ECG at Screening or Baseline (based on average of triplicate ECGs). A history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
* Left bundle branch block at Screening or Baseline
* Persistent systolic blood pressure (BP) greater than 160 or less than 100 millimeters of mercury (mmHg) or diastolic BP greater than 100 or less than 50 mmHg at Screening or Baseline
* Persistent pulse rate less than 50 beats/minute (min) or more than 90 beats/min at Screening or Baseline
* History of myocardial infarction, ischemic heart disease, or cardiac failure at Screening
* History of clinically significant arrhythmia or uncontrolled arrhythmia
* Known history of clinically significant drug allergy at Screening or Baseline
* Participants with any contraindications to diltiazem Extended Release
* Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
* Known to be human immunodeficiency virus (HIV) positive at Screening
* Active viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
* History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug or alcohol test at Screening or Baseline
* Participants who smoke or have used tobacco or nicotine-containing products within 4 weeks prior to first dose
* A Columbia Suicide Severity Rating Scale (C-SSRS) suicidal ideation score of 4 or 5 at Screening or Baseline, or for the period within 6 months before Screening or Baseline, or any lifetime suicidal behavior
* Currently enrolled in another clinical trial or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) preceding informed consent
* Engagement in strenuous exercise within 2 weeks prior to first dose (e.g., marathon runners, weight lifters)
* Intake of caffeinated beverages or caffeinated food within 72 hours prior to first dose
* Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard], and charbroiled meats) within 1 week prior to first dose
* Intake of herbal preparations containing St. John's Wort within 4 weeks prior to first dose
* Intake of over-the-counter (OTC) medications within 14 days (or 5 half-lives, whichever is longer) before dosing unless the Principal Investigator and sponsor medical monitor consider that they do not compromise participant safety or study assessments
* Use of any prescription drugs within 4 weeks prior to first dose

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with any adverse event (AE) and any serious adverse event (SAE) | up to Day 27
Mean values for the indicated hematology and blood chemistry parameters at the indicated time points | Screening; Baseline; Day 6; Day 11; Follow-up/Early Termination (FU/ET) (Day 27); Unscheduled Visits
Mean urine values at the indicated time points | Screening; Baseline; Day 6; Day 11; FU/ET (Day 27); Unscheduled Visits
Mean values for the indicated vital signs at the indicated time points | Screening; Baseline; Days 1-6; Days 12-25; FU/ET (Day 27); Unscheduled Visits
  Day 1: predose; 2, 4, 6, 8, and 12 hours postdose. Day 2: 24 hours postdose. Day 12: predose; 2, 4, 6, 8, and 12 hours postdose; Day 13: 24 hours postdose)
Mean values for the indicated electrocardiogram (ECG) parameters at the indicated time points | Screening; Baseline; Days 1-6; Days 12-25; FU/ET (Day 27); Unscheduled Visits
  Day 1: predose; 2, 4, 6, 8, and 12 hours postdose. Day 2: 24 hours postdose. Day 12: predose; 2, 4, 6, 8, and 12 hours postdose. Day 13: 24 hours postdose
Mean values for the indicted physical examination parameters at the indicated time points | Screening; Baseline; Day 11; Day 25; FU/ET (Day 27); Unscheduled Visits
Mean maximum drug concentration (Cmax) for E2027 and metabolites at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose
Mean area under the concentration x time curve from time zero to time 144 hours measurable concentration postdose (AUC[0-144]) for E2027 and metabolites at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose
Mean area under the concentration x time curve from time zero to time infinity postdose (AUC[0-inf]) for E2027 and metabolites at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose

SECONDARY OUTCOMES:
Mean area under the concentration x time curve from time zero to time 72 hours measurable concentration postdose (AUC[0-72]) for E2027 and metabolites at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose
Mean time to reach maximum (peak) concentration (tmax) for E2027 and metabolites at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose
Mean terminal elimination half-life (t1/2) for E2027 and metabolites at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose
Mean apparent total body clearance after oral administration (CL/F) for E2027 at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose
Mean apparent volume of distribution in the terminal phase (Vz/F) for E2027 at Day 1 and Day 12 | Days 1 and 12: predose; 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes